CLINICAL TRIAL: NCT05944094
Title: Evaluation of the Efficacy of Chlorhexidine Use During the First Trimester as a Regulator of Vaginal Microbiota in Reducing Preterm Birth
Brief Title: Preterm Labor Prevention Using Vaginal Antiseptics Prior to 16 Weeks of Gestation
Acronym: PLUVA
Status: Completed | Type: Observational
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Hospital Universitario La Fe (Other)
Responsible Party: Sponsor
Other Study IDs: PLUVA
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Preterm Birth
Keywords: Preterm birth, chlorhexidine, primary prevention
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Group 1: exposed patients: Group 1: pregnant women who received intravaginal chlorhexidine before 16 weeks of gestation Group 2: pregnant women who did not received intravaginal chlorhexidine e before 16 weeks of gestation
  Interventions: Device: Clorhexidine

INTERVENTIONS:
Device: Clorhexidine — Antiseptic treatment aimed at reducing potential bacterial overgrowth consisted of 10 days (1 box) of vaginal ovules of CLX (CumLaude CLX ® , CLX digluconate 0.2%) always starting between 10+0 and 16+0 weeks.
  Other Names: Code GMDN (Global Medical Device Nomenclature): 47673 - Vaginal mucosa suppository Code NBOG (Notified Body Operations Group): MD0303- CumLaude CLX ®

SUMMARY:
The aim of this prospective observational study was to evaluate the efficacy of a universal strategy of primary prevention of preterm birth using intravaginal chlorhexidine (CLX) applied before 16 weeks.

The main question is whether universal treatment with vaginal CLX before 16 weeks would reduce the incidence of preterm birth, especially before 34 weeks.

Participants were recruited at the routine first trimester consultation. All patients underwent an initial ultrasound examination between 6+0 and 15+6 weeks gestation, including assessment of embryo/fetus vitality.

Antiseptic treatment aimed at reducing possible bacterial overgrowth consisted of 10 days (1 box) of CLX vaginal ovules (CLX digluconate 0.2%) always starting between 9+0 and 16+0 weeks.

As this product is widely marketed and frequently indicated in gynaecology, we did not deprive the non-treated group of treatment because we wanted to assess whether it could have an effect on reducing preterm delivery.

The pregnant women were then followed up until the end of pregnancy and compared with a cohort of patients who had not received any treatment.

All data related to delivery were collected, as well as any events related to preterm delivery, such as onset of contractions, cervical shortening and premature rupture of membranes, regardless of final gestational age at delivery.

DETAILED DESCRIPTION:
Clinical implications of the study:

The clinical implications of our project would be to counteract the effect of pathogenic bacteria from the beginning of pregnancy (outside the teratogenic period) with the administration of the CLX ovules and thus enhance the action of the normal vaginal microbiota in the pregnant patient, since the glycogen available due to hormonal action favours the growth and development of lactobacillus, responsible for its protective activity against pathogens during pregnancy.

Sample size:

The approximate number of births per year in Spain is 370,000. The minimum number of patients to be recruited would be 400 with a 95% confidence interval.

Patients were recruited as they attended the consultation where the PI and/or collaborators were present.

Variables:

* maternal age,
* parity,
* Gestational age (GA) at examination in weeks,
* GA at delivery in weeks,
* Interval between ultrasound and delivery,
* Birth weight (BW), BW centile,
* fetal gender,
* onset of labor (elective cesarean section, induction of labor and spontaneous onset of labor),
* mode of delivery (cesarean section for abnormal cardiotocography, failure to progress or elective, assisted delivery and spontaneous delivery),
* Apgar scores at 5 minutes,
* neonatal cord arterial hydrogen potential( pH)
* Newborn destination: ward, neonatal, neonatal intensive care unit
* Type of event triggering preterm birth:Premature rupture of membranes /Uterine dynamics + cervical modifications

Statistical analysis Continuous variables were presented as mean and standard deviations (SD), median and interquartile range (IQR), while categorical variables were presented as absolute numbers and relative frequencies. Characteristics between both cohorts were compared by mean of Mann- Whitney and Fisher tests. Finally, to assess the validity of results and ensure consistency an additional multivariable analysis was performed adjusting for clinical parameters, to evaluate the odds ratio (OR) of the different determinants in the prediction of preterm birth. Finally, preterm birth incidence was calculated for specific groups selected according to the multivariable analysis result. Statistical analysis and graphs were done using Graph Pad Prism®, Mac version 9.0.1, and Stat Plus® Mac Pro version 8.0.1.s. Permissions were obtained from La Fe hospital review board and from the Valencian Autonomic Government health authorities (reference: PLUVA, date 4-2-2021). Written informed consent was retrieved to participate in the study. The authors report no conflicts of interest.

Quality control:

All analyses were performed on a single sample of patients who met the selection criteria and who had all the information required for the variables to be analysed.

In cases where it was not possible to obtain this information, the following were excluded from the study

ELIGIBILITY:
Inclusion Criteria:- Healthy pregnant patients from the 9 weeks until 15weeks 6 days who attend the first trimester check-up

Exclusion Criteria:

Patients with a history of previous preterm birth.

* Patients with vaginal bleeding during the first trimester.
* Patients with abnormalities detected in the first trimester ultrasound scan.
* Twin pregnancies
* Patients with a known allergy to the topical use of Chlorhexidine in any of its forms of presentation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population was defined by all pregnant patients previously dated by crown-rump length, who attended the initial control or first trimester screening without evident risk of preterm birth at the time of consultation at the Hospital Universitari i Politécnic La Fe during the year 2021.
Sampling Method: Probability Sample
Enrollment: 1117 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Preterm birth | 9 months
  Vaginal delivery before 34 weeks

SECONDARY OUTCOMES:
Cervical shortening | 9 months
  Cervical shortening below 25 mm before 34 weeks
Threatened preterm labor | 9 months
  presence of regular uterine contractions associated with cervical modifications (dilatation and/or shortening of the cervix) before 37 weeks
Premature rupture of membranes | 9 months
  Premature rupture of membranes before 37 weeks

CONTACTS AND LOCATIONS:
Overall Officials: José Morales-Roselló, Prof.Dr, Principal Investigator — Instituto de Investigación Sanitaria La Fe
Locations (1):
- Hospital Uiversitario y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown RG, Marchesi JR, Lee YS, Smith A, Lehne B, Kindinger LM, Terzidou V, Holmes E, Nicholson JK, Bennett PR, MacIntyre DA. Vaginal dysbiosis increases risk of preterm fetal membrane rupture, neonatal sepsis and is exacerbated by erythromycin. BMC Med. 2018 Jan 24;16(1):9. doi: 10.1186/s12916-017-0999-x. PMID 29361936
- [Result] MacIntyre DA, Chandiramani M, Lee YS, Kindinger L, Smith A, Angelopoulos N, Lehne B, Arulkumaran S, Brown R, Teoh TG, Holmes E, Nicoholson JK, Marchesi JR, Bennett PR. The vaginal microbiome during pregnancy and the postpartum period in a European population. Sci Rep. 2015 Mar 11;5:8988. doi: 10.1038/srep08988. PMID 25758319
- [Result] Romero R, Hassan SS, Gajer P, Tarca AL, Fadrosh DW, Nikita L, Galuppi M, Lamont RF, Chaemsaithong P, Miranda J, Chaiworapongsa T, Ravel J. The composition and stability of the vaginal microbiota of normal pregnant women is different from that of non-pregnant women. Microbiome. 2014 Feb 3;2(1):4. doi: 10.1186/2049-2618-2-4. PMID 24484853
- [Result] Spear GT, French AL, Gilbert D, Zariffard MR, Mirmonsef P, Sullivan TH, Spear WW, Landay A, Micci S, Lee BH, Hamaker BR. Human alpha-amylase present in lower-genital-tract mucosal fluid processes glycogen to support vaginal colonization by Lactobacillus. J Infect Dis. 2014 Oct 1;210(7):1019-28. doi: 10.1093/infdis/jiu231. Epub 2014 Apr 15. PMID 24737800
- [Result] Leitich H, Kiss H. Asymptomatic bacterial vaginosis and intermediate flora as risk factors for adverse pregnancy outcome. Best Pract Res Clin Obstet Gynaecol. 2007 Jun;21(3):375-90. doi: 10.1016/j.bpobgyn.2006.12.005. Epub 2007 Jan 22. PMID 17241817

DOCUMENTS (1):
  • Informed Consent Form (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT05944094/ICF_000.pdf